CLINICAL TRIAL: NCT00346944
Title: Health Effects From Removal of Amalgam Restorations in Patients With Symptoms Allegedly Related to Dental Amalgam - A Study of Patients Examined at the Dental Biomaterials Adverse Reaction Unit in 1993 to 1999
Brief Title: Health Effects From Removal of Amalgam Restorations in Patients With Symptoms Allegedly Related to Dental Amalgam
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Bergen (Other)
Collaborators: NORCE Norwegian Research Centre AS (Other)
Responsible Party: Principal Investigator, Lars Bjorkman, Principal Researcher, NORCE Norwegian Research Centre AS
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: REK III 24.01
Record Dates: First submitted 2006-06-29; First posted 2006-07-04 (Estimated); Last update posted 2012-08-28 (Estimated); Status verified 2012-08

CONDITIONS: Adverse Effects; Dental Restoration, Permanent

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment group (Experimental)
  Interventions: Procedure: Removal of dental amalgam restorations
- Reference group (No Intervention)

INTERVENTIONS:
Procedure: Removal of dental amalgam restorations — Removal of dental amalgam restorations by patient's own dentist. Fillings will be replaced with e.g. resin based filling material, metalloceramic restorations, and ceramic materials. Rubber dam will be used during removal of amalgam restorations.
  Arms: Treatment group

SUMMARY:
The aim of the project is to study changes in symptom load after removal of all dental amalgam restorations in patients with symptoms allegedly related to amalgam.

DETAILED DESCRIPTION:
Patients referred from dentists and physicians in the period 1993 to 1999 to the Dental Biomaterials Adverse Reaction Unit, Department of Health, UNIFOB AS, for symptoms related to amalgam restorations are randomized into treatment group (n=20) or reference group (n=20). All patients in the treatment group are followed 3, 12, 36 and 60 months after completion of amalgam removal with questionnaires on health outcomes, Minnesota Multiphasic Personality Inventory-2 (MMPI-2) and laboratory tests.

ELIGIBILITY:
Inclusion Criteria:

* Referred for examination of general health complaints related to amalgam
* Health complaints from at least three different organ systems
* Dental amalgam restorations present
* Data available on concentration of mercury in blood and urine at the initial examination
* Patient agreed to be contacted after the examination

Exclusion Criteria:

* Serious disease (incl. severe allergy to foodstuff and severe rheumatoid arthritis)
* Mental instability or psychiatric disease
* Cases with complicated dental rehabilitation (incl. bridge prostheses)
* Allergy to dental replacement materials
* Severe periodontitis
* High caries activity

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2002-09; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Changes of subjective health complaints | Five years
Changes over time of the MMPI-profile | Five years
Quality of life improvement | Five years

SECONDARY OUTCOMES:
Reduction of mercury in blood serum | One year

CONTACTS AND LOCATIONS:
Overall Officials: Lars Björkman, DDS, PhD, Principal Investigator — University of Bergen
Locations (1):
- UNIFOB AS, Dental Biomaterials Adverse Reaction Unit, Bergen, Norway

REFERENCES:
- [Background] Björkman L, Dalen K, Helland V. Clinical trial on health effects from removal of amalgam restorations. J Dent Res 84(Spec Iss A): 1192, 2005.
- [Result] Sjursen TT, Lygre GB, Dalen K, Helland V, Laegreid T, Svahn J, Lundekvam BF, Bjorkman L. Changes in health complaints after removal of amalgam fillings. J Oral Rehabil. 2011 Nov;38(11):835-48. doi: 10.1111/j.1365-2842.2011.02223.x. Epub 2011 Apr 23. PMID 21517933
- [Result] Lygre GB, Sjursen TT, Svahn J, Helland V, Lundekvam BF, Dalen K, Bjorkman L. Characterization of health complaints before and after removal of amalgam fillings--3-year follow-up. Acta Odontol Scand. 2013 May-Jul;71(3-4):560-9. doi: 10.3109/00016357.2012.697577. Epub 2012 Jul 2. PMID 22746255
- [Result] Bjorkman L, Brokstad KA, Moen K, Jonsson R. Minor changes in serum levels of cytokines after removal of amalgam restorations. Toxicol Lett. 2012 Jun 1;211(2):120-5. doi: 10.1016/j.toxlet.2012.03.769. Epub 2012 Mar 28. PMID 22475563